CLINICAL TRIAL: NCT06006325
Title: Electroacupuncture Modulates the Metabolism of SPMs and Ameliorates Respiratory Symptoms and Inflammation in Patients With Sepsis Complicating ARDS
Brief Title: Electroacupuncture Modulates SPMs Metabolism and Respiratory Symptoms in Patients With Sepsis Complicating ARDS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Nankai Hospital (Other)
Responsible Party: Principal Investigator, Jianbo Yu, Prof., Tianjin Nankai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NKYY_YXKT_IRB_2022_023_01
Record Dates: First submitted 2023-08-16; First posted 2023-08-23 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Sepsis; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Sepsis; Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture (EA) (Experimental): The acupoints were "Deqi", and the electroacupuncture stimulator was connected and energized.
  Interventions: Device: electroacupuncture treatment
- Sham electroacupuncture (SHAM-EA) (Sham Comparator): No "Deqi" operation was performed on non-acupuncture points, and the electroacupuncture stimulator was connected and not energized.
  Interventions: Device: sham electroacupuncture treatment

INTERVENTIONS:
Device: electroacupuncture treatment — Patients received acupuncture on both sides of the Zusanli (ST36) acupuncture points, and after "Deqi ", the needle was connected to an electro-acupuncture device (Hwato, Suzhou Medical ). The EA stimulation lasted for 30 min.
  Arms: Electroacupuncture (EA)
Device: sham electroacupuncture treatment — The participants in the SHAM-EA group performed shallow punctures at the bilateral non-acupuncture points, did not perform the "Deqi" operation, and were connected to the electroacupuncture stimulator but not energized.
  Arms: Sham electroacupuncture (SHAM-EA)

SUMMARY:
In this interventional clinical trial, researchers will administer electroacupuncture versus sham electroacupuncture to sepsis patients with ARDS and collect objective outcome measures. The study will be divided into 2 groups. The EA group will receive electroacupuncture and the SHAM-EA group will receive sham electroacupuncture. The purpose of this study is to investigate the effect of electroacupuncture on the synthesis of SPMs in sepsis patients with ARDS.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females over the age of 18;
2. Diagnosis meets SPESIS 3 criteria for sepsis;
3. The diagnosis meets the Berlin diagnostic criteria for ARDS;
4. ARDS was diagnosed within 48h;
5. Capable of understanding the purpose and risk of the study;
6. Patients or proxy must give written informed consent before any assessment is performed.

Exclusion Criteria:

1. ARDS was diagnosed 48h later;
2. Pregnancy, lactation or perinatal period;
3. malignant tumor;
4. Severe liver failure or kidney failure;
5. Predicted mortality risk of patients within 24h>80%;
6. Severe end-stage lung disease;
7. ECMO patients are undergoing implementation;
8. HIV seropositive or Syphilis seropositive;
9. Any clinical-relevant condition that might affect study participation and/or study results;
10. Participation in any other intervention trial;
11. Unwillingness or inability to following the study protocol in the investigators opinion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-08-20 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-10-02 (Estimated)

PRIMARY OUTCOMES:
Serum levels of Lipoxin A4 (LXA4) | Up to 7 days
  Serum levels of LXA4 were measured in post-intervention patients and levels were compared to Day 0.

SECONDARY OUTCOMES:
LXA4 levels in BALF | Up to 7 days
  LXA4 levels were measured in the BALF of patients after the intervention and the levels were compared to day 0.
Ventilation-free days | Up to 28 days
  The number of days the patient was alive and free of mechanical ventilation (MV)
Oxygenation index | Up to 7 days
  The ratio of arterial oxygen partial pressure (PaO2 in mmHg) to fractional inspired oxygen (FiO2 expressed as a fraction, not a percentage).
Ventilator-provided positive end-expiratory pressure (PEEP) | Up to 7 days
  Ventilator parameter
plateau pressure | Up to 7 days
  Ventilator parameter
tidal volume | Up to 7 days
  Ventilator parameter
Inflammation biomarkers Inflammation levels | Up to 7 days
  Procalcitonin (PCT), C-reactive protein (CRP), tumor necrosis factor-alpha (TNF-alpha), interleukin-1 beta (IL-1β), and interleukin-6 (IL-6)
Sequential Organ-Failure Assessment (SOFA) score | Up to 7 days
  The SOFA score is used to assess the severity and prognosis of sepsis.SOFA was based on six different scores, one for each of the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems each scored from 0 to 4 with an increasing score reflecting worsening organ dysfunction.
Rate of electroacupuncture-related adverse events | Up to 28 days
  Rate of electroacupuncture-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jianbo Yu, MD, Study Director — Tianjin Nankai Hospital
Locations (1):
- Tianjin Nankai Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu S, Wang Z, Su Y, Qi L, Yang W, Fu M, Jing X, Wang Y, Ma Q. A neuroanatomical basis for electroacupuncture to drive the vagal-adrenal axis. Nature. 2021 Oct;598(7882):641-645. doi: 10.1038/s41586-021-04001-4. Epub 2021 Oct 13. PMID 34646018
- [Background] Faix JD. Biomarkers of sepsis. Crit Rev Clin Lab Sci. 2013 Jan-Feb;50(1):23-36. doi: 10.3109/10408363.2013.764490. PMID 23480440
- [Background] Cecconi M, Evans L, Levy M, Rhodes A. Sepsis and septic shock. Lancet. 2018 Jul 7;392(10141):75-87. doi: 10.1016/S0140-6736(18)30696-2. Epub 2018 Jun 21. PMID 29937192
- [Background] Fowler AA 3rd, Truwit JD, Hite RD, Morris PE, DeWilde C, Priday A, Fisher B, Thacker LR 2nd, Natarajan R, Brophy DF, Sculthorpe R, Nanchal R, Syed A, Sturgill J, Martin GS, Sevransky J, Kashiouris M, Hamman S, Egan KF, Hastings A, Spencer W, Tench S, Mehkri O, Bindas J, Duggal A, Graf J, Zellner S, Yanny L, McPolin C, Hollrith T, Kramer D, Ojielo C, Damm T, Cassity E, Wieliczko A, Halquist M. Effect of Vitamin C Infusion on Organ Failure and Biomarkers of Inflammation and Vascular Injury in Patients With Sepsis and Severe Acute Respiratory Failure: The CITRIS-ALI Randomized Clinical Trial. JAMA. 2019 Oct 1;322(13):1261-1270. doi: 10.1001/jama.2019.11825. PMID 31573637